CLINICAL TRIAL: NCT01611337
Title: Insight in Persons Presenting Schizophrenia or Related Troubles During Hospitalization in Psychiatry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Esquirol (Other)
Responsible Party: Principal Investigator, Danielle Bourlot, MD, Head of Esquirol Hospital Medical Council, Centre Hospitalier Esquirol
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012-A00155-38
Record Dates: First submitted 2012-05-29; First posted 2012-06-04 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Schizophrenia
Keywords: schizophrenia, insight
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- insight evaluation (Other): insight evaluation using the Q8 scale
  Interventions: Other: insight variation measure

INTERVENTIONS:
Other: insight variation measure — insight variation between the firt week of hospitalization and 1 month later

SUMMARY:
Therapeutic alliance, and drug observance are major difficulties in the care of persons presenting schizophrenic symptomatology. They appear to be linked to insight, the consciousness that one has of his troubles. Nurse care in psychiatry aims at improving it, but usually without using specific evaluation tool. Insight is usually not evaluated during care, and its evolution is also not known, although it is highly probable that a positive evolution of insight for a person in hospital correlated to an adapted and optimal care by the medical and nursing teams. The investigators do not know examples of insight evaluation during a sequence of hospital care, or any evidence of insight variation in relation to evolution abilities of some schizophrenic patients cared in hospital.

The investigators propose here to evaluate insight in people presenting schizophrenia or related troubles, at the beginning of hospitalization (I1) and 1 month later (I2), to better characterize insight variations, and identify the sociodemographic, clinical and therapeutic variables linked to it.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia,
* Persons requiring psychiatric care in one of the participating care unit
* I1 < 6 (absent or bad consciousness of the trouble).

Exclusion Criteria:

* I1≥6
* Expression capacities incompatible with Q8 scale quotation (delirium, no understanding of the french language, mutism, contention or therapeutic isolation)
* Age under 18, absence of health care insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2012-06; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
number of collected data explaining insight variation between the first week of hospitalization (I1) and 1 month later (I2) in a model of logistic regression | first month after hospitalization
  identification of the variables explaining insight variation when it is ≥ 1,5: social and demographic data : age, gender, marital status, study level clinical : disease duration, Positive and Negative Syndrome Scale (PANSS), type of trouble therapeutic : care and treatments received during hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Bourlot, MD, Principal Investigator — Centre Hospitalier Esquirol
Locations (2):
- France (2):
  - Centre Hospitalier Esquirol, Limoges
  - Centre Hospitalier La Vallette, Saint-Vaury